CLINICAL TRIAL: NCT03943225
Title: What we Think About the Do-not-resuscitate Order: Survey Study
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Yadigar Yılmaz, anesthesiologist, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: 10840098-604.01.01-E.15467
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-05

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: The do-not-resuscitate order, end of life, medical ethics
MeSH Terms: conditions — Behavior; Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The do not resuscitate (DNR) order is a decision taken by the patient or other people about medical care in the end stages of life to withhold CPR in event of respiratory or cardiac arrest and allow natural death to occur. There is currently no related article of law to DNR order in Turkey. It was aimed to evaluate the health workers(HW) and the non health workers'(NHW) knowledge, attitude, and behavior related to the do-not-resuscitate (DNR) order in Turkey.

DETAILED DESCRIPTION:
The do not resuscitate (DNR) order is a decision taken by the patient or other people about medical care in the end stages of life to withhold CPR in event of respiratory or cardiac arrest and allow natural death to occur. There is currently no related article of law to DNR order in Turkey. A questionnaire with 25 questions has been distributed to health workers and non-health workers.

It was aimed to evaluate the health workers(HW) and the non health workers'(NHW) knowledge, attitude, and behavior related to the do-not-resuscitate (DNR) order in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* People who are able to complete the questionnaire

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health workers and non health workers who are able to complete the questionnaire
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Health workers' and Non-health workers' knowledge about the DNR order | 20-30 minutes.
  Rate of DNR order's knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Yadigar Yılmaz, Principal Investigator — Sultan Abdulhami̇d Han Eği̇ti̇m Ve Araşti̇rma Hastanesi̇
Locations (1):
- Yadigar Yılmaz, Istanbul, Turkey (Türkiye)